CLINICAL TRIAL: NCT05482087
Title: A Phase II, Multi-center, Open-label, Single-Arm Study to Evaluate the Efficacy and Safety of Oral XZP-3621 Treatment for Chinese Patients With ALK-Positive Non-Small Cell Lung Cancer
Brief Title: A Study of XZP-3621 in Chinese Patients With ALK Positive NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3621-2001
Record Dates: First submitted 2022-07-21; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: ALK-positive NSCLC
Keywords: XZP-3621; ALK-positive NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XZP-3621 (Experimental): XZP-3621 single agent,500 mg oral tables，QD，continuously
  Interventions: Drug: XZP-3621

INTERVENTIONS:
Drug: XZP-3621 — ALK inhibitor-treated ALK-positive NSCLC treatment

SUMMARY:
This was a single-arm, open-label, multicenter, phase II study to evaluate the efficacy and safety of the ALK inhibitor XZP-3621 when used as single agent in patients with ALK-rearranged stage IIIB, IIIC or IV NSCLC previously treated with other ALK inhibitors or non-previously treated.

DETAILED DESCRIPTION:
This is a Phase 2, China only, multi center, open label, three cohorts study, in ALK positive locally advanced or metastatic NSCLC patients will be enrolled to receive XZP-3621 monotherapy.

(in Cohort 1) Treatment-Naive with any ALK inhibitor. (in Cohort 2) Disease progression after crizotinib as the only ALK inhibitor. (in Cohort 3) Disease progression after other ALK inhibitors,including or not including crizotinib previously treated.

The patients will receive XZP-3621 at 500 mg orally once daily (QD), taken with food.Patients will be treated until disease progression, unacceptable toxicity, withdrawal of consent, or death, whichever occurred first. After disease progression (as per RECIST v1.1), patients should discontinue the study medication. After disease progression, patients will be treated at the discretion of the investigator according to local practice. Information regarding the nature and the duration of subsequent therapies will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18-75 years-of-age;
2. Patients with Histologically or cytologically confirmed diagnosis of advanced or recurrent (Stage IIIB and IIIC not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC that is ALK-positive where ALK status is determined by Ventana immunohistochemistry (IHC) test or FISH or PCR or NGS,Sufficient tumor tissue available to perform ALK status is required if not determined.
3. Subject should have:

   (in Cohort 1) Treatment-Naive with any ALK inhibitor. (in Cohort 2) Disease progression after crizotinib as the only ALK inhibitor. (in Cohort 3) Disease progression after other ALK inhibitors,including or not including crizotinib previously treated.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 2;
5. All Subjects must have at least 1 measurable extracranial target lesion according to RECIST v1.1 that has not been previously irradiated.
6. CNS metastases are allowed if:

   1. Asymptomatic: either untreated and not currently requiring corticosteroid treatment, or
   2. Previously diagnosed and treatment has been completed with full recovery from the acute effects of radiation therapy or surgery prior to enrollment, and if corticosteroid treatment for these metastases has been withdrawn for at least 4 weeks with neurological stability.
   3. Such cases are not be allowed,such as leptomeningeal disease (LMD) or carcinomatous meningitis (CM) if visualized on magnetic resonance imaging (MRI), or if baseline CSF positive cytology is available .
7. Have recovered from toxicities related to prior anticancer therapy to national cancer institute common terminology criteria for adverse events (NCI CTCAE) v5.0 grade less than or equal to (<=)2. (Note: treatment-related alopecia and AEs that in the investigator's judgment do not constitute a safety risk for the subject are allowed.)
8. Prior chemotherapy and radiotherapy (other than palliative) must be completed at least 4 weeks prior to initial administration; Palliative radiotherapy must be completed 1 week prior to initial administration.
9. Patients treated with any ALK inhibitor must be discontinued for ≥5 half-life or 14 days, whichever is longer, before XZP-3621 tablets are first administered;
10. Life expectancy of at least 12 weeks;
11. Adequate organ system function, defined as follows:

    1. Absolute neutrophil count (ANC) ≥1.5 x 109/L; Platelets ≥100 x 109/L;Hemoglobin ≥9 g/dL (≥90 g/L)
    2. Total bilirubin ≤1.5 times the upper limit of normal (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 *ULN if no liver involvement or ≤5 * ULN with liver involvement.
    3. Creatinine < 1.5 *ULN. If >1.5 * ULN, patient may still be eligible if calculated creatinine clearance >50 mL/min (0.83mL/s) as calculated by the Cockcroft-Gault method.
12. Serum pregnancy test (for females of childbearing potential) negative at screening.
13. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

  1. Combined with small cell lung cancer;
  2. Uncontrolled malignant pleural/peritoneal effusion and/or pericardial effusion (uncontrolled means that the effusion increases significantly within one week after extraction and has obvious symptoms requiring further puncture or other intervention) ;
  3. Patients with a previous malignancy within the past 5 years are excluded (other than curatively treated basal cell carcinoma of the skin, early gastrointestinal (GI) cancer by endoscopic resection, in situ carcinoma of the cervix.);
  4. Previous treatment history of organ transplantation, hematopoietic stem cell or bone marrow transplantation;
  5. Patient has had major surgery within 4 weeks prior (2 weeks for resection of brain metastases) to the first dose of study drug or has not recovered from side effects of such procedure;
  6. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C virus (HCV) (eg, in case of known HBsAg or HCV antibody positivity);
  7. Known human immunodeficiency virus (HIV);
  8. Clinically active infections affecting the safety of subjects, including active tuberculosis;
  9. Uncontrolled hyperglycemia;
  10. Subject with predisposing characteristics for acute pancreatitis according to investigator judgment, including but not limited to current gallstone disease,history of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease within 28 days of initial administration;
  11. Subject with uncontrolled electrolyte disturbances (e.g., low calcium, low magnesium, or hypokalemia) that are identified by investigator;
  12. Unable to swallow;
  13. History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis;
  14. Clinically significant vascular (both arterial and venous) and non-vascular cardiac conditions, (active or within 3 months prior to enrollment), which may include, but are not limited to:

      1. Arterial disease such as cerebral vascular accident/stroke (including Transient Ischemic Attack -TIA), myocardial infarction, unstable angina;
      2. Venous diseases such as cerebral venous thrombosis, symptomatic pulmonary embolism;
      3. Non-vascular cardiac disease such as congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree AV block (unless paced) or any AV block with PR >220 msec; or ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, etc.), machine-read Electrocardiogram (ECG) with QTc >470 msec, or congenital long QT syndrome;
  15. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 150 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 95 mm Hg;
  16. Patient has impairment of GI function or GI disease that may significantly alter the absorption of XZP-3621 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome);
  17. Patient receiving treatment with medications that meet one of the following criteria and that cannot be discontinued at least 14 days prior to the start of treatment with XZP-3621 and for the duration of the study;

      * Strong inhibitors or strong inducers of CYP3A4.
      * Medications with a known risk of prolonging the QT interval or inducing Torsades de Pointes.
  18. Participation in other studies involving investigational drug(s) within 28 days prior to study entry and/or during study participation;
  19. Pregnant female patients; breastfeeding female patients;
  20. History of hypersensitivity to any of the additives in the XZP-3621 or crizotinib drug formulation;
  21. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior;
  22. laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator and/or the sponsor, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-05-07 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | From Cycle 1 Day 1 to documented progression of disease by Investigator (up to 20 months)[Note:Each cycle is 28 days]..
  ORR was defined as the proportion of patients with a best overall response defined as Complete Response (CR) or Partial Response (PR) as evaluated by investigator assessment per RECIST 1.1.CR was defined as the disappearance of all target lesions. PR was defined as a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | From Cycle1 Day1 to the date of the first documented disease progression(up to overall period of approximately 20 months)[Note:Each cycle is 28 days]..
  PFS was defined as the time (in months) from first dose to the first documentation of disease progression, as Determined by Investigator Using RECISTv1.1., or to death from any cause, whichever occurred first.
Overall Survival (OS) | From Cycle 1 Day 1 until death (up to approximately 20 months)[Note:Each cycle is 28 days]..
  OS was defined as the time from date of first dose to date of death due to any cause,as Determined by the investigator Using RECISTv1.1.
Duration of Response (DoR) | From first documentation of CR or PR to documented progression of disease by Investigator( up to approximately 20 months)
  DoR defined as the time from date of first documented CR or PR to date of first documented disease progression or death due to any cause,whichever occurred first.
Disease Control Rate (DCR) | Baseline, Week 8, thereafter every 8 weeks until disease progression, death or withdrawal from the study (up to overall period of approximately 20 months)
  DCR defined as the proportion of patients with best overall response of CR, PR, or Stable Disease (SD).
Intracranial Objective Response Rate(IC-ORR) | From Cycle 1 Day 1 to documented progression of disease by Investigator (up to 20 months).
  Intracranial objective response rate(IC-ORR) was defined as the same as ORR (defined as the percentage of participants with a best overall confirmed response of CR or PR according to RECIST version 1.1 relative to the total participants in the analysis population), but limited to Intra Cranial lesions only on participants with central nervous system metastases.
Area Under the Plasma Concentration-time Curve (AUC) of XZP-3621 and Its Metabolite | Predose and 4 hours post dose on Day 1 of Cycle1;Predose on Day15 of Cycle1; Predose on Day1 of Cycle2,Cycle3 and Cycle4(each cycle is 28 days);
  AUC was collected for both XZP-3621 and its major metabolite, and was based on their concentrations in plasma over time.
Maximum Plasma Concentration Observed (Cmax) of XZP-3621 and Its Metabolite | Predose and 4 hours post dose on Day 1 of Cycle1;Predose on Day15 of Cycle1; Predose on Day1 of Cycle2,Cycle3 and Cycle4(each cycle is 28 days);
  Cmax was collected for both XZP-3621 and its major metabolite, and was based on their concentrations in plasma over time.
Percentage of Participants With Non-serious Adverse Events and Serious Adverse Events | From Screening (within 28 days prior to Cycle 1 Day 1) through and including at least 30 days after the last administration of the investigational product, up to 23 months(each cycle is 28 days).
  Percentage of Participants With Non-serious Adverse Events and Serious Adverse Events. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, MD, Principal Investigator — Jilin Province Cancer Hospital
Locations (1):
- Jilin Province Cancer Hospital, Jilin, Chang Chun, China